CLINICAL TRIAL: NCT01688674
Title: Dextrose Boluses Versus Dextrose Infusions by Burettes in Prevention of Hypoglycemia Among Preterms Admitted at Mulago Hospital: An Open Label Randomized Clinical Trial
Brief Title: Dextrose Infusion by Burettes Versus Dextrose Boluses in Prevention of Neonatal Hypoglycemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was more benefit from the infusion arm compared to the bolus arm.
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, KUTAMBA ELIZABETH, Elizabeth Kutamba.R, Makerere University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009/HD11/16712 U
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Once a Preterm Developed Hypoglycemia, no More Blood Glucose Was Measured During the Study Period.
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bolus arm (Placebo Comparator): two hourly dextrose boluses administered via an intravenous cannula
  Interventions: Drug: 10% dextrose
- infusion (Experimental): 10% dextrose infusion by burettes
  Interventions: Drug: 10% dextrose

INTERVENTIONS:
Drug: 10% dextrose

SUMMARY:
NULL HYPOTHESIS • There is no difference in the incidence of hypoglycemia among preterms receiving either two hourly 10% dextrose boluses or 10% dextrose infusion by burettes during the 72 hours of admission in Special Care Unit- Mulago Hospital.

ALTERNATE HYPOTHESIS

• Use of two hourly 10% dextrose boluses increases the incidence of hypoglycemia by 30% compared to 10% dextrose infusion by burettes among preterms admitted to Special Care Unit in the first 72 hours of admission.

ELIGIBILITY:
Inclusion Criteria:

- SELECTION CRITERIA Inclusion criteria

* Preterms whose care givers/ mothers gave informed consent
* Preterms whose age was < 24 hours of life
* Preterms with birth weight ≥1kg
* Preterms with random blood sugar ≥ 2.6 mmol/l at admission into SCU.

Exclusion Criteria

* Absence of a biological mother or abandoned baby
* Presence of gross congenital abnormalities.
* Very sick (Apgar score ≤ 5 at 5 minutes

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence proportion of hypoglycemia | 3months

SECONDARY OUTCOMES:
survival measured as a proportion | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago Hospital, Kampala, Mulago, Uganda

REFERENCES:
- [Derived] Kutamba E, Lubega S, Mugalu J, Ouma J, Mupere E. Dextrose boluses versus burette dextrose infusions in prevention of hypoglycemia among preterms admitted at Mulago Hospital: an open label randomized clinical trial. Afr Health Sci. 2014 Sep;14(3):502-9. doi: 10.4314/ahs.v14i3.2. PMID 25352865